CLINICAL TRIAL: NCT00702052
Title: An Open-Label, Single-Arm, Phase II Study of RAD001 in Patients With Mantle Cell Lymphoma Who Are Refractory or Intolerant to Velcade® (Bortezomib)
Brief Title: Safety and Efficacy of RAD001 in Participants With Mantle Cell Lymphoma Who Are Refractory or Intolerant to Velcade® Therapy
Acronym: PILLAR-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001N2201; 2007-005700-40 (EudraCT Number)
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Results first posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-04

CONDITIONS: Lymphoma, Mantle- Cell
Keywords: Mantle Cell Lymphoma; Lymphoma; B-Cell Lymphoma; Mantle Zone Lymphoma; Refractory Lymphoma; Aggressive Lymphoma; PILLAR-1
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma; Lymphoma, B-Cell | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Everolimus (Experimental): Participants received everolimus tablets, 10 mg, orally, once daily during each 28 day cycle until determination of objective tumor progression or unacceptable toxicity, or death, or consent withdrawal, or discontinuation from the study for any other reason.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Everolimus tablets
  Other Names: RAD001

SUMMARY:
This study was to evaluate the safety and efficacy of a daily, oral dose of 10 mg RAD001 in participants with Mantle Cell Lymphoma who were refractory or intolerant to Velcade® therapy and who had received at least one prior antineoplastic agent other than Velcade®, either separately or in combination with Velcade® (see inclusion criteria). Intolerance to Velcade® therapy was determined by the study investigator based on clinical evaluations. Participants were considered refractory to Velcade® if they have documented radiological progression on or within 12 months of the last dose of Velcade® when given alone or, on or within 12 months of the last dose of the last component of a combination therapy which included Velcade®.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (≥18 years old) with Mantle Cell Lymphoma that has been confirmed by central pathology review (archival diagnostic tumor specimen required).
* Participants with mantle cell lymphoma who have documented refractory disease to Velcade® (bortezomib) or who have documented intolerance to Velcade® therapy. Intolerance to Velcade® is determined by the study investigator based on clinical evaluations. Participants are considered refractory to Velcade® if they have documented radiological progression on or within 12 months of last dose of Velcade® when given alone or, on or within 12 months from the last dose of the last component of a combination therapy which included Velcade®. Participants are considered refractory to Velcade®, if Velcade® is part of a combination treatment for the disease.
* Participants must have received at least one prior antineoplastic agent, other than Velcade® either separately or in combination with Velcade® (bortezomib).
* At least one site of measurable nodal disease at baseline >2.0 cm in the longest transverse diameter and clearly measurable in at least two perpendicular dimensions, as determined by computer tomography (CT) scan (or magnetic resonance imaging (MRI), only if CT scan can not be performed).
* Eastern Cooperative Oncology Group (ECOG) performance status = 0, 1 or 2.
* Life expectancy ≥3 months.
* Adequate bone marrow, liver and renal function.
* Platelets ≥75 x 10^9/L (untransfused platelets).

Exclusion Criteria:

* Participants who are currently receiving anticancer therapies or have received anticancer therapies within 4 weeks of the start of study drug (including chemotherapy, radiation, antibodies, targeted therapy etc.) are not eligible.
* Previous treatment with mammalian target of rapamycin (mTOR) inhibitors (e.g. everolimus, sirolimus, temsirolimus, etc).
* Participants with prior allogeneic stem cell transplant.
* Grade 3 or 4 unresolved toxicity from prior antineoplastic therapies.
* Currently taking other investigational agents or received other investigational drugs within 4 weeks of the start of study drug.
* Participants with central nervous system (CNS) lymphoma are not eligible; head magnetic resonance imaging (MRI) (or computer tomography (CT) if MRI is not available) is required prior to study entry.
* Use of chronic, systemic corticosteroids or another immunosuppressive agent, except prednisone ≤20 mg daily (or equivalent) for adrenal insufficiency (must have been on a stable dosage regimen for ≥4 weeks prior to the first treatment with RAD001).
* HIV positive participants are not eligible; (human immunodeficiency virus (HIV) testing is not required for study entry; review of previous medical records is required).
* Uncontrolled hyperlipidemia (≥Grade 3 hyperlipidemia despite optimal supportive medical therapy).
* Active, bleeding disorders or major surgery within 4 weeks of starting study drug.
* Severe and/or uncontrolled medical conditions such as symptomatic congestive heart failure (New York Heart Association Class III or IV), unstable angina, myocardial infarction within 6 months or study start, severely impaired lung function, cirrhosis, chronic active/persistent hepatitis.
* History of another primary malignancy ≤3 years prior to study entry.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-08-22 (Actual); Primary Completion 2012-04-20 (Actual); Study Completion 2012-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (31):
- United States (31):
  - Mayo Clinic - Arizona Mayo Clinic - Scottsdale, Multiple Locations, Arizona
  - Highlands Oncology Group DeptofHighlandsOncologyGrp(2), Fayetteville, Arkansas
  - Bay Area Cancer Research Dept.ofBayAreaCancerResearch, Concord, California
  - City of Hope National Medical Center Dept.ofCityofHopeMedicalCtr(1), Duarte, California
  - UCLA/ University of California Los Angeles Dept.of Hem/Oncology, Los Angeles, California
  - University of California Davis Cancer Center Dept. of UC Davis Cancer (4), Sacramento, California
  - Rocky Mountain Cancer Centers RMCC - Denver-Midtown, Greenwood Village, Colorado
  - Advanced Medical Specialties Medical Onc Hem, Miami, Florida
  - Georgia Health Sciences University Dept. of MCG, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - St. Francis Cancer Research Foundation Dept.ofSt.FrancisCancerRes.(2), Beech Grove, Indiana
  - Central Indiana Cancer Centers CICC - East (2), Indianapolis, Indiana
  - University of Michigan Comprehensive Cancer Center Dept of Michigan Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic - Rochester Hematology, Rochester, Minnesota
  - Washington University School Of Medicine-Siteman Cancer Ctr Medical Oncology, St Louis, Missouri
  - Hackensack University Medical Center Dept ofHackensackUniversityMC, Hackensack, New Jersey
  - New York University Medical Center NYU Cancer Institute, New York, New York
  - East Carolina University BrodySchool of Medicine, Greenville, North Carolina
  - Northwest Cancer Specialists Vancouver Cancer Center (2), Portland, Oregon
  - Kaiser Permanente Northwest Dept of Kaiser Northwest (3), Portland, Oregon
  - Fox Chase Cancer Center Regulatory Contact, Philadelphia, Pennsylvania
  - Western Pennsylvania Cancer Institute /Western Penn Hospital Western Pann. Cancer Inst., Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center Hillman Cancer Center (4), Pittsburgh, Pennsylvania
  - Cancer Centers of the Carolinas CC of C -Eastside, Greenville, South Carolina
  - Vanderbilt University Medical Center, Clinical Trials Center Dept. of VUMC, Nashville, Tennessee
  - Baylor College of Medicine Dept. of Sammons Cancer (2), Dallas, Texas
  - University of Texas Southwestern Medical Center DeptofSimmons Cancer Center(2), Dallas, Texas
  - MD Anderson Cancer Center/University of Texas Dept. of MD Anderson (10), Houston, Texas
  - Tyler Cancer Center Dept.ofTylerCancerCtr., Tyler, Texas
  - Cancer Care Northwest CC Northwest- Spokane South(3), Spokane, Washington
  - West Virginia University/ Mary Babb Randolph Cancer Center, Morgantown, West Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 26 investigative sites in the United States from 22 August 2008 to 20 April 2012.
Period: Overall Study
Arm/Group | Everolimus
Started | 58
Completed | 0
Not Completed | 58
Not completed — Adverse Event | 23
Not completed — Disease Progression | 30
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all participants who received at least one dose of the study drug.
Arm/Group | Everolimus
Number analyzed (Participants) | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.29 (7.991)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 45

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate was defined as the percentage of participants with a best overall disease response of complete response (CR) or partial response (PR). CR was defined as complete disappearance of all extranodal lesions. PR was defined as at least a 50% decrease in the sum of the product of diameter (SPD) of all index nodal and extranodal lesions.
Time Frame: From date of enrollment up to disease progression or death (approximately 3.8 years)
Population: The Full Analysis Set (FAS) included all participants who received at least one dose of the study drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Everolimus
Number analyzed (Participants) | 58
percentage of participants | 8.6 [3.5 to 17.3]

2. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease Control Rate was defined as the percentage of participants with best overall disease response of CR or PR or stable disease (SD). CR was defined as complete disappearance of all extranodal lesions. PR was defined as at least a 50% decrease in SPD of all index nodal and extranodal lesions. SD was defined failure to attain the criteria needed for CR or PR and failure to fulfill the criteria for at least a 50% increase in the SPD of all index nodal and extranodal (including splenic and/or hepatic nodules) lesions, taking as reference the smallest sum of the product of the diameters of all index lesions recorded at or after baseline.
Time Frame: From date of start of treatment up to disease progression or death (approximately up to 3.8 years)
Population: The FAS included all participants who received at least one dose of the study drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Everolimus
Number analyzed (Participants) | 58
percentage of participants | 69.0 [57.5 to 78.9]

3. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from the date of first documented disease response (CR or PR) to the date of first documented progression or death due to lymphoma. CR was defined as complete disappearance of all extranodal lesions. PR was defined as at least a 50% decrease in SPD of all index nodal and extranodal lesions.
Time Frame: From date of start of treatment up to disease progression or death (approximately up to 3.8 years)
Population: We have exhausted all efforts to locate this data and it has since been destroyed, therefore no data is available to report for this outcome measure.
Arm/Group | Everolimus
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of start of treatment to the date of event defined as the first documented progression or death due to any cause.
Time Frame: From date of start of treatment up to disease progression or death (approximately up to 3.8 years)
Population: The FAS included all participants who received at least one dose of the study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus
Number analyzed (Participants) | 58
months | 4.40 [3.48 to 6.08]

5. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of start of study treatment to the date of death due to any cause.
Time Frame: From date of start of treatment up to disease progression or death (approximately up to 3.8 years)
Population: The FAS included all participants who received at least one dose of the study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus
Number analyzed (Participants) | 58
months | 16.85 [14.36 to 29.86]

6. Secondary Outcome: Number of Participants With At Least One Adverse Event (AE) and Serious Adverse Event (SAE)
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. A SAE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important.
Time Frame: From the start of the study and 28 days after study drug discontinuation (approximately up to 18 months)
Population: The safety set included all participants who received at least one dose of the study drug with a valid post-baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 58
Participants
  AE | 58
  SAE | 29

ADVERSE EVENTS:
Time Frame: From the start of the study and 28 days after study drug discontinuation (approximately up to 18 months)
Description: The safety set included all participants who received at least one dose of the study drug with a valid post-baseline assessment.
Arm/Group | Everolimus
All-Cause Mortality (participants affected / at risk) | 7/58
Serious Adverse Events (participants affected / at risk) | 29/58
Other Adverse Events (participants affected / at risk) | 58/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=58)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Intracardiac thrombus (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Multi-organ failure (General disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Arthritis infective (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Clostridial infection (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 6
Sinusitis (Infections and infestations) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=58)
Anaemia (Blood and lymphatic system disorders) | 15
Leukopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 17
Tachycardia (Cardiac disorders) | 4
Lacrimation increased (Eye disorders) | 4
Vision blurred (Eye disorders) | 6
Abdominal distension (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 11
Constipation (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 26
Dry mouth (Gastrointestinal disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Haemorrhoids (Gastrointestinal disorders) | 5
Mouth ulceration (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 16
Oral pain (Gastrointestinal disorders) | 4
Proctalgia (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 12
Toothache (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 10
Asthenia (General disorders) | 8
Fatigue (General disorders) | 25
Oedema peripheral (General disorders) | 16
Pain (General disorders) | 4
Pyrexia (General disorders) | 12
Bronchitis (Infections and infestations) | 3
Candidiasis (Infections and infestations) | 3
Herpes zoster (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 5
Sinusitis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 7
Urinary tract infection (Infections and infestations) | 4
Aspartate aminotransferase increased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 3
Blood triglycerides increased (Investigations) | 4
Platelet count decreased (Investigations) | 4
Weight decreased (Investigations) | 8
Decreased appetite (Metabolism and nutrition disorders) | 13
Dehydration (Metabolism and nutrition disorders) | 5
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 8
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hyponatraemia (Metabolism and nutrition disorders) | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Dizziness (Nervous system disorders) | 9
Dysgeusia (Nervous system disorders) | 8
Headache (Nervous system disorders) | 11
Hypoaesthesia (Nervous system disorders) | 3
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Blister (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e. data from all sites) in the clinical trial.